CLINICAL TRIAL: NCT01665040
Title: Precision Spectra™ Neurostimulator System for the Treatment of Chronic Intractable Pain of the Trunk and/or Limbs
Brief Title: Clinical Outcomes Study Using a New Implantable Neurostimulation System for Chronic Intractable Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5004
Record Dates: First submitted 2012-08-09; First posted 2012-08-15 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain
Keywords: neurostimulation; spinal cord stimulation; peripheral nerve stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neurostimulation for chronic pain (Experimental): Neurostimulation (spinal cord stimulation with or without peripheral nerve stimulation of the trunk) for chronic intractable pain of the trunk and/or limbs.
  Interventions: Device: Neurostimulation device implantation

INTERVENTIONS:
Device: Neurostimulation device implantation — Study subjects will undergo a screening-trial of neurostimulation using the Boston Scientific Corporation Precision Spectra neurostimulation system and may proceed to permanent implantation in the event of a successful screening trial.
  Treatment will include spinal cord stimulation and may also include peripheral nerve stimulation, based upon the physician's subject-specific treatment plan.

SUMMARY:
The primary objective of this study is to investigate patient satisfaction with treatment using a new implantable neurostimulation system for chronic pain of the trunk and/or limbs.

ELIGIBILITY:
Inclusion Criteria:

* Chronic intractable pain of the trunk and/or limbs
* Documented history of trunk and/or limb pain of at least 180 days
* Overall pain intensity of at least 5 on a 0-10 numerical rating scale (OPI-NRS-11) over the past 180 days based on subject recall
* Pass study site's routine psychological/psychiatric evaluation within 180 days before signing the informed consent
* Subject is willing and able to comply with all protocol-required follow-up evaluations
* 18 years of age or older when written informed consent is obtained
* Subject signs informed consent

Exclusion Criteria:

* Unable to operate the Precision Spectra™ System either by self or with a caregiver
* Primary source of pain is cancer-related, pelvic, visceral, anginal or migraine
* Overall pain intensity of always 10 on a 0-10 numerical rating scale (OPI-NRS-11) over the past 180 days based on subject recall
* Is a high surgical risk
* Currently on any anticoagulant medications that cannot be discontinued during perioperative period
* Subject requires Magnetic Resonance Imaging (MRI) while implanted with lead(s) and/or the Precision Spectra IPG
* Subject is participating (or intends to participate) in another investigational drug or device clinical trial that may influence the data that will be collected for this study
* Subjects already implanted with an active implantable device(s) to treat their pain (IPGs, implantable drug pumps, etc) or pacemaker or Implantable Cardiac Defibrillator
* Patient is a woman who is pregnant (a urine pregnancy test must be performed within 7 days prior to the stimulation trial procedure in women of child-bearing potential) or nursing or intends to become pregnant during the course of the trial.
* Failed to achieve satisfactory relief during the stimulation trial phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Neuromodulation Corporation
Locations (7):
- Australia (2):
  - Metro Spinal Clinic, Caulfield
  - Hunter Clinical Research, Melbourne
- AZ Delta, Roeselare, Belgium
- Spain (4):
  - Clinica Universitaria de Navarra, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Quiron Madrid, Madrid
  - H. Clinico Universitario, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Neurostimulation for Chronic Pain: Neurostimulation (spinal cord stimulation with or without peripheral nerve stimulation of the trunk) for chronic intractable pain of the trunk and/or limbs.
  Neurostimulation device implantation: Study subjects will undergo a screening-trial of neurostimulation using the Boston Scientific Corporation Precision Spectra neurostimulation system and may proceed to permanent implantation in the event of a successful screening trial.
  Treatment will include spinal cord stimulation and may also include peripheral nerve stimulation, based upon the physician's subject-specific treatment plan.
Period: Overall Study
Arm/Group | Neurostimulation for Chronic Pain
Started | 40
Completed | 36
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Neurostimulation for Chronic Pain
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Satisfied With Treatment at 90 Days Post-IPG Implantation
Description: Proportion of subjects satisfied with treatment at 90 days post-IPG implantation, as measured by a 7-point Patient Satisfaction with Treatment (PSWT) questionnaire.
Time Frame: 90-days post permanent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Neurostimulation for Chronic Pain
Number analyzed (Participants) | 40
Participants | 32

2. Primary Outcome: Proportion of Subjects Satisfied With Treatment in a Sub-group Utilizing More Than 2 IPG Ports at 365 Days Post-IPG Implantation
Description: Proportion of subjects in a sub-group utilizing more than 2 IPG ports at 365 Days post-IPG implantation satisfied with treatment, as measured by a 7-point Patient Satisfaction with Treatment (PSWT) questionnaire.
Time Frame: 365 days post permanent implantation
Population: A sub-group of subjects utilizing more than 2 IPG ports at 365 Days post-IPG implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Neurostimulation for Chronic Pain
Number analyzed (Participants) | 21
Participants | 21

ADVERSE EVENTS:
Time Frame: 365 days
Description: The investigator was responsible for notifying the IRB/IEC of deviations from the CIP, serious adverse events (SAEs) or unanticipated adverse device effects (UADEs) occurring at the site, and other SAE/UADE reports received from the Sponsor (BSC) in accordance with local procedures and IRB/IEC requirements.
Arm/Group | Neurostimulation for Chronic Pain
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 11/40
Other Adverse Events (participants affected / at risk) | 4/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurostimulation for Chronic Pain (N=40)
Infection (Infections and infestations) | 5 (5)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 3 (4)
Nervous System Disorders (Nervous system disorders) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurostimulation for Chronic Pain (N=40)
Falls (Injury, poisoning and procedural complications) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes